CLINICAL TRIAL: NCT02712762
Title: Dry Eye and Ocular Surface Disease in Chronic Graft-Versus-Host Disease (GVHD) Patients
Brief Title: Ocular Surface Disease in Chronic Graft-Versus-Host Disease (GVHD) Patients
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Louis Tong, Principal Investigator, Singapore National Eye Centre
Other Study IDs: R1312/118/2015; 2016/2085 (Registry Identifier: SingHealth CIRB)
Record Dates: First submitted 2016-03-08; First posted 2016-03-18 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Dry Eye; GVHD
Keywords: immunological profiles
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cross-sectional study

SUMMARY:
This study aims to profile the ocular surface inflammation of chronic Graft-Versus-Host Disease patients by investigating conjunctival cells, and clinical imaging for conjunctival redness and tear stability. Hence, the investigators expect to find an increased in inflammatory cell population in GVHD conjunctival samples.

DETAILED DESCRIPTION:
Dry eye is a multi-factorial disease that is frequently encountered in ophthalmological practice. Common dry eye symptoms include eye irritation, heaviness of the eyelids, blurred vision and light sensitivity (1). The worldwide prevalence of dry eye is generally high (2-4). In Asia, dry eye may affect up to 22% of adults above 40 years in China (5) and Japan (3). In Asian patients older than 65 years, prevalence rates of dry eye can be as high as 80% if diagnosis is based on abnormal tear stability, or as high as 60% on meibomian gland dysfunction (MGD), a major cause of tear instability (6).

Most dry eye patients can be successfully managed with lubricants, punctal occlusion, steroid and/or cyclosporine eye drops. However, some patients with severe dry eye and likely underlying diseases for example Graft-Versus-Host Disease (GVHD), who have exhausted conventional treatments may amount to 10-20 cases a year and are difficult to manage. These patients and their physicians are helpless when faced with these scenarios.

Hematopoietic stem cell transplantation (SCT) has been established as a potential curative therapy for hematologic malignancies (9). The number of SCT recipients has increased exponentially worldwide over the past 2 decades. GVHD is the major cause of morbidity and mortality in patients undergoing allogeneic SCT (10).

Dry eye associated with chronic GVHD is one of the major late complications after allogeneic SCT; it has a significant impact on patients' quality of life (11-13) and can lead to blindness (14). The immunological process of dry eye associated with chronic GVHD remains largely unknown but is believed to be traditional alloreactivity to recipient tissues.

The investigators propose to collaborate with Singapore General Hospital, Department of Haematology to focus on the clinical characteristics and immunological profile of the ocular surface inflammation in more severe chronic GVHD patients. Dry eye severity is more severe in chronic GVHD patients at SNEC, compared to idiopathic cases of dry eye. This may be due to referral bias, or may be related to the systemic disease. As such, the investigators intend to do a pilot study to define some ocular characteristics of non-referred haematology patients with GVHD. The investigators propose to screen and recruit 30 suitable participants who have chronic GVHD. Tests to be performed will include ocular imaging (Oculus K5M), ocular immunological profile (conjunctiva immune cells) and ocular surface inflammation (MMP-9 tear marker).

1 HYPOTHESIS AND OBJECTIVES

This study thus aims to profile the ocular surface inflammation of chronic GVHD patients by investigating conjunctival cells, and clinical imaging for conjunctival redness and tear stability. Hence, the investigators expect to find an increased in inflammatory cell population in GVHD conjunctival samples.

Specific aims:

1. To determine the ocular immunological profile (conjunctival immune cells) of patients with GVHD and correlate to systemic status (treatment).
2. To determine if objective measures of tear dysfunction/ ocular surface inflammation are abnormal in GVHD patients, and correlate to systemic status.

Outcomes:

* Dry eye symptoms (SPEED Questionnaire)
* Tear production
* Conjunctival immune cells profile (Proportion of T lymphocytes and other immune cells)
* Clinical parameters for ocular surface (conjunctival redness, non-invasive tear break-up time, corneal fluorescein staining)

Long term aims:

1. To establish criteria for screening cGVH patients for referral to ophthalmic specialists.
2. To determine longitudinal outcomes of cGVH dry eye cases, and effects of systemic prophylactic treatment, as well as other ocular treatment such as plasmapheresis eye drops.

1.1.1 Potential Risks The investigators will anticipate minimal risk and discomfort involve in this study.

* It is possible that there may be some slight discomfort during the sampling of conjunctival cells using the impression membrane
* Some slight discomfort from tear Strip Meniscometry
* Participants may feel slight irritation when the InflammaDry test kit is administered, as it requires placing a soft pad made of absorbent material on the participant's lower lid to collect tears.
* Stinging sensation as a result of local anaesthetic (Alcaine)

1.1.2 Potential Benefits With greater understanding of the presence of various inflammatory mediators, the investigators can gain further insight into the complex process taking place in chronic GVHD patients.

2 STUDY POPULATION 3.1 List The Number and Nature of Subjects to be Enrolled. Thirty eligible GVHD patients will be screened and recruited from Transplant Centre located at Block 7, Level 1, Singapore General Hospital- Department of Haematology.

3.2 Criteria for Recruitment and Recruitment Process

1. Subjects meet all the inclusion criteria
2. Clear of exclusion criteria.

Permission would be sought from the attending doctors from SGH, Department of Haematology before subjects are being recruited. Eligible subjects will be counselled on the study. If subject is interested, informed written consent will be obtained from all participants. After which, SERI research optometrist will proceed with ocular examination at SGH Transplant Centre.

4 STUDY DESIGN

4.1.1 Study Procedures

The examinations will be done by SERI study team members. The list of required examinations is shown:

1. Dry Eye Symptoms (SPEED Questionnaire)
2. Non-invasive Tear Break-up Time (NIKBUT)- Oculus K5M
3. Conjunctival Redness- Oculus K5M
4. Tear Strip Meniscometry (SMTube), Schirmers test
5. Tear MMP-9 result (Inflammadry)
6. Impression Cytology- using EyePrim conjunctival membranes
7. Corneal Fluorescein Staining- Oculus K5M

Details of procedures

1. Dry Eye Questionnaire Participants will be asked to score dry eye questionnaire to assess the symptomatic severity of dry eyes and the extent of its disruption to daily activities for the past two weeks.

   • SPEED Questionnaire Consist of 2 questions on frequency and severity graded on a scale of 0-3 on frequency and grade 0-4 on severity. The questionnaire allows patient to rate from 0 which is never and 3 which is all the time in frequency and 0 as no problem and 4 as intolerable in severity.
2. Non Invasive Tear Break-up Time (NIBUT) The Oculus keratographer 5M (Oculus, Wetzlar, Germany) will be used to perform the non-invasive tear break up time. Patient will sit comfortably in front of the instrument and blink freely while fixing on a target directly ahead. Once the patient is ready, patient will be instructed to blink twice and refrain from blinking. Keratograph 5M is fully automated and it will capture any break or distortion in the image and the time of the break will be noted. Three readings will be taken for each eye to get the average value. It is possible that the tear film of participants is more stable, i.e. increased tear break up time.
3. Imaging of conjunctival redness with Oculus Keratography 5M
4. Tear Strip Meniscometry (SMTube) Remove SMTube from the sterile pouch. Hold the centre of SMTube. Do not touch the dye area. Immerse the tip of the SMTube to the lateral lower lid tear meniscus of an eye for 5 seconds. Take extra precaution to prevent the tip from touching the patients' conjunctiva. After 5 seconds, remove the SMTube from the lower lid tear meniscus. Measure the length of the column stained blue in colour.
5. Tear MMP-9 result (Inflammadry) The InflammaDry test will be administered after tear meniscometry is performed, as it assesses the MMP-9 levels (an inflammatory marker) in tears and hence is not affected by reflex tearing (15). The fleece of the test strip is dab along the inside lining of the lower eyelid in multiple locations, the patient is asked to blink, and the strip is then rest along the inferior nasal palpebral conjunctival for another 5 seconds. Assemble the sampling fleece into the sample transfer window of the test cassette body. After which the absorbent tip is immersed in the buffer solution for 20 seconds. Remove the absorbent tip from the buffer vial, replace the protective cap, and lay the test flat on the horizontal surface for 10 minutes. A single blue line indicates a negative result, while the appearance of 2 lines (red and blue) indicates a positive result.
6. Impression Cytology (using EyePrim membranes)

   i) Preparation of RPMI solution In a sterile biosafety hood, prepare 2 vials of 2ml Eppendorf tubes. One tube for right eye and left eyes respectively. Fill the 2 tubes with 1.5ml of RPMI solution. Thereafter, transfer tubes in ice-box containing ice and transfer to the Transplant Centre located at SGH where impression will be done.

   ii) Anaesthesia Step 1: Inform the participant that he/she may experience a transient stinging sensation. Request for the participant to direct their gaze upwards. Depress the lower eyelid and place one drop of LA in the inferior palpebral fornix. Do this for both eyes. Request for the patient to blink gently for at least 3 times. Step 2: Once the stinging subsides, request for the participant to direct their gaze downwards. Elevate the patient's upper eyelid and place a drop of LA on the bulbar conjunctiva on the most superior point possible. Do this for both eyes. Request for the patient to blink gently for at least 3 times. Step 3: Repeat step 2 once more. The participant should not be able to feel any stinging sensations of the eye at this point.

   iii) Conjunctival sampling Step 1: Request the participant to direct his/her gaze in the infero-temporal direction. This exposes the superior nasal bulbar conjunctiva for impression. Step 2: Apply the EyePRIM membrane to the area. Step 3: Ensure good apposition of the membrane with the conjunctiva. Do this by rocking the EyePRIM membrane to the left and right. Step 4: Remove the membrane from the conjunctiva with a peeling-like movement. Step 5: Exert greater force on the EyePRIM spring mechanism. After a "click" sound, the membrane will be ejected from the gadget. Place the membrane from the right eye into the "right" eppendorf tube. Step 6: Repeat for the superior temporal bulbar conjunctiva, this time directing the participant's gaze infero-nasally. Place this membrane into the "right" eppendorf tube. There should be 2 membranes in this eppendorf tube. Step 7: Place this tube in the box of ice. Step 8: Repeat steps 1-7 for the other eye, but place the membranes into the "left" eppendorf tube. Step 9: At this point should have both "right" and "left" eppendorf tubes, each with 2 membranes within them immersed in 1.5ml of RPMI medium. Place them in the ice box.

   iv) Detachment of cells from membranes Using a 10ul micropipette tip, scrape the cells off the membrane. Ensure to scrape the correct side of the membrane (this can be done by referring to the direction of the hooks of the membrane). This is most easily done by pinning down the membrane against the wall of the vial tube and scraping it off with a grinding-like motion (the wall of the vial tube is the mortar and the micropipette tip is like a pestle). Repeat for the other membrane in the same vial tube. Also, repeat the same steps for the other eye. Once scraping of cells is completed, placed the 2 eppendorf tubes onto the ice and hand over to the Aihua or Tanima (Academia Level 12) for FACs analysis on the same day.
7. Corneal fluorescein staining score

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed with chronic Graft Versus Host Disease (GVHD).

Exclusion Criteria:

1. No ocular surgery within the last 3 months and LASIK within 1 year.
2. Ocular surface diseases such as pterygium, or obvious lid/orbital disease with lagophthalmos.
3. Any other specified reason as determined by clinical investigator.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a cross-sectional study involving 30 consecutive suitable GVHD patients. Suitable patients will be identified by haematologists from the SGH transplantation Centre (Block 7, level 1).
  Study duration: One visit
  Recruitment duration: 1 Year
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-06; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Dry Eye Symptoms (SPEED Questionnaire) | Baseline

SECONDARY OUTCOMES:
Non-invasive Tear Break-up Time (NIKBUT) | Baseline
Imaging of Conjunctival Redness | Baseline
  These parameters will be imaged and measured by Keratograph 5M. Briefly, the participant will be asked to look at a target in the instrument while blinking normally. The keratographer will scan the ocular surface and images will be captured. The grading of the conjunctival hyperemia will be automatically performed relative to standard pictures of increasing redness stored on the system.
Tear production with Schirmers I test | Baseline
  This will be done with the standard Schirmer Tear Test Strips from Clement Clark currently used at SERI (5 mm wide with a notch for folding). No prior anaesthetic will be used. The strips will be positioned over the inferior temporal half of the lower lid margin in both eyes at the same time. Subjects will be asked to close their eyes. Any excessive irritation signs will be noted. The extent of the wetting in each strip will be recorded after 5 minutes of testing. The strip will be collected and stored in 1.5 ml eppendorf tubes at -80˚C until further analysis.
Measuring tear biomarker | Baseline
Conjunctival Immune Cell Profile | Baseline
  Proportions of T lymphocytes and other immune cells
Corneal Fluorescein Staining Score | Baseline
  A drop of normal saline will be instilled on the fluorescein strip (Fluorets) then shaken off so that no visible drop remains. The subject is asked to look up before the introduction of the fluoret to the inferior conjunctival fornix on the right then left eye. Corneal fluorescein staining will be imaged by Keratograph 5M. Scoring system will be based on CCLRU. Briefly, there will be 5 corneal zones. The staining scale is 0-4, with 0.5 unit steps in each of the zones.

CONTACTS AND LOCATIONS:
Locations (1):
- Cynthia Boo, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No